CLINICAL TRIAL: NCT05195541
Title: A Clinical Study to Evaluate the Safety, Pharmacokinetic Profile and Efficacy of CU-20401 Administered Subcutaneously in the Submental Fat (SMF) Population
Brief Title: A Clinical Study to Evaluate the Safety, Pharmacokinetic Profile and Efficacy of CU-20401
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CU-20401-104
Record Dates: First submitted 2021-12-02; First posted 2022-01-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Safety
Keywords: pharmacokinetic profile; efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort A1 (Experimental): 0.02mg/injection，2 injections
  Interventions: Drug: CU-20401
- Cohort A2 (Experimental): 0.04mg/injection，2 injections
  Interventions: Drug: CU-20401
- Cohort B1 (Experimental): 0.04mg/injection，4 injections
  Interventions: Drug: CU-20401
- Cohort B2 (Experimental): 0.075mg/injection，4 injections
  Interventions: Drug: CU-20401
- Cohort C1 (Experimental): 0.075mg/injection，6 injections
  Interventions: Drug: CU-20401
- Cohort C2 (Experimental): 0.15mg/injection，6 injections
  Interventions: Drug: CU-20401
- cohort X1 (Experimental): 0.04mg/injection，20 injections
  Interventions: Drug: CU-20401
- cohort X2 (Experimental): 0.075mg/injection，20 injections
  Interventions: Drug: CU-20401
- cohort X3 (Experimental): 0.15mg/injection，20 injections
  Interventions: Drug: CU-20401
- cohort X (Placebo Comparator): 0.15mg of placebo /injection，20 injections
  Interventions: Drug: CU-20401

INTERVENTIONS:
Drug: CU-20401 — Subcutaneous injection in the subcutaneous fat area，0.2ml
  Other Names: injection，CU-20401

SUMMARY:
This study is a Phase Ib/II clinical study. Phase 1b was a single-center, nonrandomized, single-arm study to evaluate the safety, PK profile, preliminary efficacy, and immunogenicity of different groups (SC) of CU-20401 in the submental fat accumulation population. Phase 2 is a multicenter, randomized, placebo parallel-controlled study to evaluate the safety, efficacy, and immunogenicity of the preferred group (SC) of CU-20401 in a submental fat accumulation population.

DETAILED DESCRIPTION:
Eligible subjects will first enter Arm A1, receive treatment for this group on D1, and undergo study visits and biological sample collection (PK samples and immunogenicity samples) at established timepoints. After the last subject in Arm A1 has completed at least 3 days of safety and tolerability observation,After no safety events (≥ Grade 2 study drug-related AEs) have occurred as assessed by the investigator, enrollment into the A2 Arm may be initiated. Enrollment in subsequent treatment groups and so on. If a subject in this dose group experiences an AE ≥ Grade 2 related to the investigational product, the investigator will assess the time to continue observation and start the next treatment group according to the subject ' s condition.

Based on the data obtained in Phase 1b, the grouping for Phase 2 will be determined by the investigator and the sponsor in consultation. It may be Group X1, Group X2, and Group X3. Eligible subjects were randomized 1: 1: 1: 1 to receive treatment in Group X1, X2, X3, or placebo on D1 and to undergo study visits and biological sample collection (immunogenicity samples) at established timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the trial contents, study process and possible adverse reactions, be able to complete the study in accordance with the protocol requirements, have reasonable expectations for the cosmetic effect of injection, and voluntarily sign the informed consent form;
2. Men or women aged 18 to 65 years (including boundary values) at screening;
3. Body mass index (BMI) was in the range of 17-40 (kg/m2) (including cut-off value) at screening;
4. At screening, the investigator assessed moderate to severe submental outline protrusion due to submental fat accumulation according to the clinician-reported Submental Fat Rating Scale (CR-SMFRS) (see Annex 1), i.e., those with a score of 2 to 3 points;
5. Non-pregnant and lactating women, and subjects (including males and females) have no pregnancy plan and voluntarily take effective contraceptive measures at screening and throughout the trial, and have no sperm or egg donation plans.

   -

Exclusion Criteria:

1. Subjects who have received prior surgery, liposuction therapy, or injection of lipolytic drugs similar to the investigational drug (e.g., phosphatidylcholine, etc.) at the submental site;
2. Those who have received biomaterial fillings (e.g., hyaluronic acid, collagen, etc.) in the neck or chin before screening;
3. Those who have received botulinum toxin injection in the neck or submental area within 3 months prior to screening, or have received noninvasive skin tightening therapy;
4. Planned to undergo cosmetic procedures at the submental site during the study, including, but not limited to, dermal filling, surgical wrinkle removal, photoelectric therapy, water light needles, microneedles, chemical peeling, or scar removal surgery, etc.;
5. Enlargement of the submental area due to other causes of excess non-submental fat accumulation (e.g., goiter, lymphadenopathy, Madelong's disease, platysma protrusion at rest, etc.) or affect the investigator's assessment of submental fat;
6. Those with obvious scars, infections, cancerous or precancerous lesions and/or unresolved wounds, retrognathia, etc. in the chin and neck position, which may affect the evaluation results as assessed by the investigator;
7. According to the investigator's judgment, submental fat dissolution can cause submental skin relaxation (SMSLG) of Grade 4 or other anatomical features (e.g., protrusion of fat under the platysma, extreme skin relaxation of the neck or submental area, protrusion of the platysma band), resulting in unacceptable cosmetic results;
8. Subjects with a pre-existing tendency to scar hyperplasia or keloid may affect the efficacy assessment or subject safety after treatment as judged by the investigator;
9. Subjects with symptoms of dysphagia or related diseases at screening;
10. Vital signs, physical examination, clinical laboratory tests (AST or ALT values above twice the upper limit of normal; serum creatinine 1.5 times higher than the upper limit of normal) and electrocardiogram at screening showed abnormalities and judged to be clinically significant, and the investigator considered it inappropriate to participate in this study;
11. Presence of other acute or chronic diseases (including but not limited to cardiovascular and cerebrovascular, respiratory, endocrine, digestive, renal, liver, blood and lymphatic, immune, metabolic and bone, central nervous system or psychiatric disorders, etc.) that may increase the risk associated with the use of the investigational product as judged by the investigator,Or may affect the interpretation of the study results, or fail to cooperate well with the trial personnel;
12. Subjects who are positive for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, treponema pallidum antibody (Anti-TP) at screening;
13. Coagulation test results (prothrombin time, partial thromboplastin time) within 4 weeks prior to dosing suggest the presence of any clinically significant bleeding disorder (subjects treated with antiplatelet therapy, anticoagulant, and acetylsalicylic acid may be enrolled after a 7-day washout period);
14. Those who have used topical medications (e.g., glucocorticoids, tretinoin ointment) in the submental region within 4 weeks prior to screening or are expected to require use in the submental area during the study (up to 12 weeks after the completion of the last injection);
15. Plan any surgery during the trial that may result in significant weight change (≥ 10%) or take any medication that may result in significant weight change (≥ 10%) (e.g. systemic corticosteroids, bariatric medications, bariatric surgery);
16. Donation of blood or massive blood loss (≥ 400 mL) within 3 months prior to screening;
17. Those with a history of needle sickness and blood sickness and significant abnormal clinical manifestations;
18. History of drug abuse within 6 months prior to screening, or drug use within 3 months prior to screening (including but not limited to morphine, methamphetamine,ketamine, tetrahydrocannabinol acid, methylenedioxymethylamphetamine, etc.);
19. Alcoholics or regular drinkers within 3 months prior to the trial, i.e., more than 21 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine), or those with a positive alcohol breath test.
20. Allergic constitution, history of allergy to collagenase or components of the study drug or its excipients;
21. Received collagenase treatment within 6 months prior to screening;
22. Participation in any drug within 3 months prior to screening or medical device clinical trials within 1 month prior to screening;
23. Lactating and pregnant women;
24. Those who cannot tolerate magnetic resonance imaging (MRI) (e.g., with a pacemaker/electronic stimulator, an insulin pump, a cochlear implant, or stainless steel metal implanted in the body, etc.);
25. Other conditions judged by the investigator to be inappropriate for participation in this study.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of local skin reactions | 1 month
  Local skin reaction(LSR）such as erythema, edema, mild tenderness, bruising, pain, and tingling/burning sensation, and other adverse events. Local skin reactions (LSR) were assessed using a 4-point scale (0 = absent at all, 1 = mild, limited involvement, 2 = moderate involvement, 3 = severe, severe involvement).
Occurrence of other adverse events | 1 month
  such as abnormalities in laboratory tests, electrocardiograms, etc

SECONDARY OUTCOMES:
Proportion of subjects with Submental Fat（SMF）Grade ≤ 1 | 1 month
  Proportion of subjects with Submental Fat（SMF）Grade ≤ 1 assessed by the investigator using Clinician-Reported Submental Fat Rating Scale（CR-SMFRS），0=absent at all，1=mild，2=moderate，3=severe，4=very severe
Changes in SMF skin laxity compared to baseline | 1 month
  The investigator assessed the change from baseline in SMF skin relaxation using Submental Skin Relaxation Scale （SLRS）.1=absent at all，2=mild，3=moderate，4=severe。
The proportion of subjects with SMF score ≥ 3 points | 1 month
  The proportion of subjects with SMF score ≥ 3 points was assessed by Subject Self-Rating Scale（SSRS), 0=very dissatisfied，1=dissatisfied，2=Generally satisfied，3=A little satisfied，4=very satisfied
Proportion of subjects with at least a 10% reduction from baseline in submental fat area | 1 month
  Proportion of subjects with at least a 10% reduction from baseline in submental fat area using MRI.
Changes in overall aesthetics compared to baseline | 1 month
  Change from baseline in Global Aesthetic Improvement Scale (GAIS) score，1=Very noticeable improvement，2=noticeable improvement，3=A little improvement，4=No improvement，5=Even worse
Changes in SMF compared to baseline | 1 month
  The investigator assessed the change from baseline in SMF skin relaxation using Patient-Reported Submental Fat Rating Scale(PR-SMFRS)，0= Fat free，1=a little fat，2=a moderate amount of fat，3=a lot of fat，4=very many fats

CONTACTS AND LOCATIONS:
Overall Officials: byron zhu', MD, Study Chair — CMO
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No